CLINICAL TRIAL: NCT05643781
Title: Tuberculosis as a Risk Factor for a Severe Course and Adverse Long-term Outcome of a Symptomatic Sars-CoV-2 Infection in Johannesburg, South Africa
Brief Title: Tuberculosis as a Risk Factor for a Worse Outcome Post-Sars-CoV-2 Infection
Acronym: Co-TB
Status: Completed | Type: Observational
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Chris Hani Baragwanath Academic Hospital (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: AUR2-8-296
Record Dates: First submitted 2022-10-20; First posted 2022-12-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Tuberculosis; Post-acute COVID-19 Syndrome
MeSH Terms: conditions — COVID-19; Tuberculosis; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum, whole blood (EDTA), PAXGene blood collected for Covid 19-serology-, inflammatory/transcriptomic- and immunology- analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Co-TB Group: Follow up all participants from hospital discharge until 12 months post-Covid-19 infection. Conduct investigations assessing cardiopulmonary, socioeconomic, quality of life outcomes. No interventions.

SUMMARY:
This study has two main objectives. First, the clinical characteristics and outcomes of hospitalized patients with symptomatic Covid-19 disease will be compared between persons with a history of past or current TB infection or disease and those, who have had no TB history. The possible impact of an HIV-coinfection will be also addressed in the planned investigations and analysis. Second, the long-term consequences and clinical outcomes of Covid-19 up to 12 months post-infection will be analysed in both groups (with and without TB history) with the main focus on cardio-pulmonary outcomes.

DETAILED DESCRIPTION:
This study is retrospective/prospective clinical observational study.

Primary Objective, Study Phase A (hospitalization, retrospective data collection):

* To describe the development and characteristics of Covid-19 pneumonia, clinically and using radiological methods (i.e. CT-thorax)
* To describe disease severity of Covid-19 disease, including treatment in Intensive Care Unit (ICU) and ventilation support measures
* To describe different types of organ failures apart from respiratory failure (e.g. kidney, liver, heart)
* To describe treatment outcomes at discharge, including cause of death
* To assess the significance of additional risk factors such as HIV infection, smoking, malnutrition, etc., for the clinical course and characteristics of a Covid-19 disease Primary Objective, Study Phase B (after end of hospitalization, prospective data collection): The primary objective of the study phase B (after end of hospitalization) is the description of Covid-19 sequelae (focus on cardio-pulmonary morbidity) in patients with and without previous TB disease during a six month follow up period after discharge from hospital, including:
* the description (characteristics and severity) of abnormal function tests and clinical examination results (e.g. in lung function measurement, cardiac tests and ECG, kidney function, neurological & mental tests)
* the definition of time to healing (ad integrum) after a Covid-19 infection
* the studying of chronic restrictions of the long-term quality of life at 12 months after discharge from hospital that are based on chronic organ failures and mental disorders
* the assessment of exacerbations of chronic organ failures, hospitalizations and deaths in 12 months phase after discharge from hospital

Secondary Objective(s):

* To collect longitudinal data that could allow for further insights on whether previous Covid-19 disease results in an increased risk for re-activation of

  /infection with M. tuberculosis
* To perform longitudinal immunological investigations in a sub-set of patients to study Covid-19- immune-activation, depending on M.tb and/or HIVcoinfection status

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide a written informed consent or witnessed oral consent in the case of illiteracy for participation in the study prior to all study-related procedures
* Be ≥ 18 years and <70 years of age
* Having a diagnosis of SARS-CoV-2 infection, confirmed by PCR tests and/or chest CT-scan
* Willing to be tested for active and latent M.tb infection and to provide information on previous TB disease episodes (including agreement for confirmation of active TB disease by the investigators, e.g. via NTP/lab registration number)
* Willing to be tested for HIV, if status is not known or the last documented negative is more than 4 weeks old
* Willingness to comply with the protocol and visit schedule, at the discretion of the investigator
* Having a firm home address that is readily accessible for visiting and is willing to inform the study team of any change of address during study participation

Exclusion Criteria:

* Has a recent history of a medical condition that is the leading cause for the current clinical symptoms and/or survival, e.g. advanced stages of cancer
* Has severe medical or psychiatric condition which in the opinion of the site investigator or designee, might interfere with the ability to give true informed consent and to adhere to the study requirements.
* Is currently imprisoned
* Confirmed or suspected pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises the general population (of 18 years and older), which is served by the study hospital. Those who cannot give informed consent, or are under imprisonment, or suffer from other medical or mental conditions and/or life under circumstances that may prevent the completion of 6 months follow up will also not be included.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Covid-19 recovery and course and the impact of tuberculosis (TB) or no tuberculosis infection. | March 2021 to December 2022
  Describe the long-term clinical characteristics and course of recovery post-Covid-19 and compare patients groups with TB infection and those without TB infection.
  TB infection will be determined by a history of TB disease, or current TB disease on medical records, and latent TB infection will be determined by Interferon-Gamma release assay blood test. Those with any positive of the above tests will be considered to have TB infection, and those with all negative tests will be considered to have no TB infection.

SECONDARY OUTCOMES:
Hospitalisation and Covid-19 severity | March 2021 to December 2022
  Describe Covid-19 pneumonia hospitalisation with Covid severity in our post-hospitalisation cohort up to 12 months post-infection.
Cardiac outcomes post-Covid-19. | March 2021 to December 2022
  Determine Covid-19 pneumonia cardiac characteristics in our post-hospitalisation cohort up to 12 months post-infection.
Lung function assessment post-Covid-19. | March 2021 to December 2022
  Describe respiratory assessment in our post-hospitalisation cohort up to 12 months post-infection.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Rachow, PhD, med, Principal Investigator — Division of Infectious Diseases and Tropical Medicine, Medical Center of the University of Munich (LMU)
Locations (1):
- The Aurum Institute, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No
Currently conducting study analysis with the database and once study is complete will discuss the plan to share IPD